CLINICAL TRIAL: NCT01160120
Title: Generic Fixed Dose Combination (FDC) of Tenofovir(TDF) /Lamivudine(3TC)/Efavirenz (EFV) Tablets 300/300/600 mg
Brief Title: Therapeutic Drug Monitoring (TDM) in Generic Tenofovir/Lamivudine/Efavirenz
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Mylan Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HIV-NAT 118
Record Dates: First submitted 2010-06-09; First posted 2010-07-12 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV
Keywords: fixed dose combinations; tenofovir; lamivudine; efavirenz; therapeutic drug levels; safety and efficacy; HIV; To evaluation new formulations of FDC of TDF/3TC/EFV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Patients can be either treatment-naïve or treatment-experienced when entering this clinical trial. After meeting the inclusion and exclusion criteria, patients will start with generic FDC of TDF/3TC/EFV 1 pill a day at night time. Only patient who are on individual TDF 3TC and EFV will undergo TDM sampling ( 11-13 hours after dosing) at baseline.
  Interventions: Drug: generic FDC of TDF/3TC/EFV

INTERVENTIONS:
Drug: generic FDC of TDF/3TC/EFV — Patients who were on individual TDF 3TC and EFV regimen before baseline will undergo TDM at baseline. Therapeutic drug monitoring (TDM) of generic FDC of TDF/3TC/EFV will be done after 4 weeks, to ensure steady state. At baseline and week 4 safety data will be obtained. In order to assess the efficacy and the long term safety of this drug, at week 12, 24 and 48 viral load, CD4 and safety parameters will be obtained.

SUMMARY:
The purpose of this study is to determine the mid levels of the tenofovir, lamivudine, and efavirenz, and 144 weeks safety and efficacy of the generic fixed dose combination of tenofovir /lamivudine/efavirenz tablets 300/300/600 mg in Thai HIV-infected patients.

DETAILED DESCRIPTION:
The trial drug FDC of TDF/3TC/EFV is a new formulation combining fixed doses of the nucleoside reverse transcriptase inhibitors lamivudine 300 mg and tenofovir disoproxil fumarate 300 mg with the non nucleoside reverse transcriptase inhibitor efavirenz 600 mg for once daily and one-tablet HAART. Co-formulated TDF/3TC/EFV demonstrated bioequivalent to original individual EFV 3TC and TDF in Indian healthy volunteers (unpublished data). It has not been evaluated in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Evidence of HIV infection
* Age> 18 years
* On a TDF/3TC/EFV (separated pills) containing HAART regimen with a VL < 50 copies within 24 weeks or ARV naïve
* eGFR >70 cc/min
* Currently having no AIDS defining illness
* No history of NRTI/NNRTI/PI failure
* Willing to adhere to the protocol requirements

Exclusion Criteria:

* Any history of taking CYP450 inhibitors or inducers drugs within 14 days of enrollment in the study
* Current pregnancy or lactating or plan to be pregnant
* Active opportunistic infection
* ALT more than 2 x upper limit
* Creatinine more than 1.5 time the upper limit
* Active drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
mid levels of TDF, 3TC, and EFV between brand and generic | 144 weeks
  mid levels of TDF, 3TC, and EFV between brand and generic

SECONDARY OUTCOMES:
kidney, liver, CD4 and viral load overtime | 144 weeks
  kidney, liver, CD4 and viral load overtime

CONTACTS AND LOCATIONS:
Overall Officials: Anchalee Avihingsanon, MD, PhD, Principal Investigator — The HIV Netherlands Australia Thailand Research Collaboration
Locations (1):
- HIV-NAT, Bangkok, Thailand

REFERENCES:
- [Result] Avihingsanon A, Sophonphan J, Thammajaruk N, Chaihong P, Burger D, Cressey TR, Ramautarsing RA, Praditornsilpa K, Avihingsanon Y, Ruxrungtham K and HIV-NAT 114 study team. Plasma Tenofovir Concentrations and Proximal Tubular Dysfunction in HIV-Infected Adults Receiving Tenofovir in Thailand. AIDS Clin Res 2015, 6:7 Doi: http://dx.doi.org/10.4172/2155-6113.1000477
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org